CLINICAL TRIAL: NCT02064361
Title: High Intensity Cycling Before SCUBA Diving Reduces Post-decompression Microparticle Production and Neutrophil Activation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Split (Other)
Collaborators: University of Maryland (Other)
Responsible Party: Principal Investigator, Zeljko Dujic, Professor Zeljko Dujic MD, PhD, University of Split
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SCUBACYC
Record Dates: First submitted 2014-02-12; First posted 2014-02-17 (Estimated); Last update posted 2014-02-17 (Estimated); Status verified 2014-02

CONDITIONS: Decompression Sickness; SCUBA Diving
Keywords: SCUBA diving; exercise,; microparticles; neutrophil activation,; high intensity exercise
MeSH Terms: conditions — Decompression Sickness; Motor Activity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- High intensity exercise (Experimental): A dive to 18 meters sea water for a duration of 41 minutes preceded by high intensity cycling
  Interventions: Other: High intensity exercise

INTERVENTIONS:
Other: High intensity exercise — Subjects performed a repeated Wingate protocol for the exercise condition of the study. This consisted of 4, 30 s maximal efforts on a weight-braked cycle ergometer (Monark 894E, Monark Exercise AB, Sweden) with 4 min active recovery between efforts, preceded by a 5 min warm up. The resistance was set at 7.5% bodyweight for the intervals and 2% for the warm up and active recovery periods.

SUMMARY:
The purpose of this study is to determine the impact of high intensity,anaerobic exercise, in the form of cycling, on SCUBA diving. Outcomes are determined by the quantification and subtype of circulating microparticles, complete blood counts, and the quantification of venous gas emboli, measured via transthoracic echocardiography, in the cardiac cavities.

ELIGIBILITY:
Inclusion Criteria:

* Experienced divers (> 250 logged dives)
* Male
* Physician clearance to dive

Exclusion Criteria:

* Prior incidence of decompression sickness

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-02; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline values of number of circulating microparticles per microliter of blood | Prior to exercise, prior to diving, 15 and 120 minutes after surfacing

CONTACTS AND LOCATIONS:
Overall Officials: Zeljko Dujic, MD. PhD, Principal Investigator — University of Split
Locations (2):
- University of Maryland, Baltimore, Maryland, United States
- University of Split School of Medicine, Split, Dalmatia, Croatia

REFERENCES:
- [Background] Thom SR, Milovanova TN, Bogush M, Yang M, Bhopale VM, Pollock NW, Ljubkovic M, Denoble P, Madden D, Lozo M, Dujic Z. Bubbles, microparticles, and neutrophil activation: changes with exercise level and breathing gas during open-water SCUBA diving. J Appl Physiol (1985). 2013 May 15;114(10):1396-405. doi: 10.1152/japplphysiol.00106.2013. Epub 2013 Mar 14. PMID 23493363